CLINICAL TRIAL: NCT05704842
Title: Pilot Study to Evaluate the Impact of a Home-Based Exercise Program on Cancer-Related Fatigue in Breast Cancer Patients Undergoing Curative-Intent Chemotherapy
Brief Title: Evaluate Impact of Exercise Program on Fatigue in Breast Cancer During Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB-2021-04
Record Dates: First submitted 2022-12-29; First posted 2023-01-30 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Other): Intervention: Subject will be assessed by a Physical Therapist. Based on the assessment, the Physical Therapist will provide the patient with a home-based exercise program including core exercises as follows: Core Stabilization, core extension, leg extensions, squats with and without weights, shoulder and arm exercises. Patients will be asked to complete a symptom survey weekly via a web-based platform for tracking cancer and treatment-related symptoms and fatigue.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Subject will not be provided an exercise program but will be asked to complete the symptom survey weekly via a web-based platform for tracking cancer and treatment-related symptoms and fatigue.

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise program including core exercises as follows: Core Stabilization, core extension, leg extensions, squats with and without weights, shoulder and arm exercises.
  Other Names: Exercise program
  Arms: Exercise

SUMMARY:
Assess feasibility of home exercise in reducing fatigue in subjects with breast cancer receiving curative intent chemotherapy. Subjects are randomized to control (no exercise) or intervention group (exercise). The PRO-CTCAE tool and FACIT Fatigue Scale are used to collect patient reported outcomes. Subjects submit data via mobile phone, tablet or computer. Assessments are weekly during chemotherapy (10-20 wks), at end of chemotherapy and 1, 3 and 6 months after chemotherapy.

DETAILED DESCRIPTION:
The goal of this project is to determine the feasibility of a specific home-based exercise intervention in reducing cancer-related fatigue (CRF) in breast cancer patients undergoing curative-intent chemotherapy. The outcome will be measured by using the FACIT Fatigue Scale, administered by using the Carevive PROmpt® platform.

Primary Objectives:

1. . To examine the feasibility of recruitment and retention of women undergoing treatment for breast cancer over the duration of the chemotherapy regimen.
2. To examine the adherence to the exercise regime for those in the intervention group and compare the retention rates between treatment and control groups
3. To compute the means and standard deviations (SD) of the FACIT responses over time in both groups for use in future power analyses to aid in the design of a futre hypothesis testing RCT.

Secondary Objectives:

1. To quantify the change over time in PRO-CTCAE derived symptoms and other PROs by computing means and SD.
2. To test for group differences in the trajectory of change over time in FACT using a Mixed Model repeated analysis

ELIGIBILITY:
Inclusion Criteria:

* Women with curative-intent breast cancer who plan to undergo at least 4 cycles of chemotherapy.
* Age > 18 years
* ECOG performance score < 3
* English-speaking
* with sufficient vision/hearing or family support
* Coronary artery disease, if cleared by cardiologist
* Subject must have smart phone, computer or tablet.
* Willingness to be randomized

Exclusion Criteria:

* Medical or psychiatric conditions (beyond those related to breast cancer and its treatment) that would impair our ability to test study hypotheses (psychotic disorders, dementia, inability to give informed consent or follow instructions).
* Patients with overt evidence of a psychiatric disorder.
* Coronary artery disease, not cleared by cardiologist.
* Contraindication to exercise.
* Chronic fatigue syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of a specific home-based exercise program in reducing cancer-related fatigue. | Baseline
  The outcome will be measured by using the FACIT Fatigue Scale 0 - 4. 0 = (not at all) 1= (a little bit) 2 = (somewhat) 3 = (Quite a bit), 4 = (Very much).
Determine the feasibility of a specific home-based exercise program in reducing cancer-related fatigue. | Weekly for 12 weeks
  Changes in fatigue will be assessed, this outcome will be measured by using the FACIT Fatigue Scale, 0 - 4. 0 = (not at all) 1= (a little bit) 2 = (somewhat) 3 = (Quite a bit), 4 = (Very much).
Determine the feasibility of a specific home-based exercise program in reducing cancer-related fatigue. | Month 1 following completion of chemotherapy
  Changes in fatigue will be assessed this outcome will be measured by using the FACIT Fatigue Scale, 0 - 4. 0 = (not at all) 1= (a little bit) 2 = (somewhat) 3 = (Quite a bit), 4 = (Very much).
Determine the feasibility of a specific home-based exercise program in reducing cancer-related fatigue. | Month 3 following completion of chemotherapy
  Changes in fatigue will be assessed, this outcome will be measured by using the FACIT Fatigue Scale, 0 - 4. 0 = (not at all) 1= (a little bit) 2 = (somewhat) 3 = (Quite a bit), 4 = (Very much).
Determine the feasibility of a specific home-based exercise program in reducing cancer-related fatigue. | Month 6 following completion of chemotherapy
  Changes in fatigue will be assessed this outcome will be measured by using the FACIT Fatigue Scale, 0 - 4. 0 = (not at all) 1= (a little bit) 2 = (somewhat) 3 = (Quite a bit), 4 = (Very much).

SECONDARY OUTCOMES:
To quantify the change over time in PRO-CTCAE derived symptoms | Baseline
  Outcome will be measured using PRO-CTCAE Derived Symptoms and other PROs. A scale Yes or No is utilized to describe whether the following symptoms have been experienced: Anxiety, constipation, decreased appetite, diarrhea, fatigue, general pain, insomnia, mouth sores, muscle pain, nausea, numbness and tingling, problems and concentration, rash, sad, shortness of breath, vomiting. The following sale: Rarely, occasionally, frequently or almost constantly will be used to measure anxiety and general pain. Severity of the following symptoms: Anxiety, fatigue, general pain and problems with concentration in a 7 day time period will be measured using the following scale: Mild, Moderate, Severe, Very Severe.
To quantify the change over time in PRO-CTCAE derived symptoms | Weekly for 12 weeks
  Changes in symptoms will be assessed this outcome will be measured using PRO-CTCAE Derived Symptoms and other PROs. A scale Yes or No is utilized to describe whether the following symptoms have been experienced: Anxiety, constipation, decreased appetite, diarrhea, fatigue, general pain, insomnia, mouth sores, muscle pain, nausea, numbness and tingling, problems and concentration, rash, sad, shortness of breath, vomiting. The following scale: Rarely, occasionally, frequently or almost constantly will be used to measure anxiety and general pain. Severity of the following symptoms: Anxiety, fatigue, general pain and problems with concentration in a 7 day time period will be measured using the following scale: Mild, Moderate, Severe, Very Severe.
To quantify the change over time in PRO-CTCAE derived symptoms | Month 1 following completion of chemotherapy
  Changes in symptoms will be assessed this outcome will be measured using PRO-CTCAE Derived Symptoms and other PROs. A scale Yes or No is utilized to describe whether the following symptoms have been experienced: Anxiety, constipation, decreased appetite, diarrhea, fatigue, general pain, insomnia, mouth sores, muscle pain, nausea, numbness and tingling, problems and concentration, rash, sad, shortness of breath, vomiting. The following scale: Rarely, occasionally, frequently or almost constantly will be used to measure anxiety and general pain. Severity of the following symptoms: Anxiety, fatigue, general pain and problems with concentration in a 7 day time period will be measured using the following scale: Mild, Moderate, Severe, Very Severe.
To quantify the change over time in PRO-CTCAE derived symptoms | Month 3 following completion of chemotherapy
  Changes in symptoms will be assessed this outcome will be measured using PRO-CTCAE Derived Symptoms and other PROs. A scale Yes or No is utilized to describe whether the following symptoms have been experienced: Anxiety, constipation, decreased appetite, diarrhea, fatigue, general pain, insomnia, mouth sores, muscle pain, nausea, numbness and tingling, problems and concentration, rash, sad, shortness of breath, vomiting. The following scale: Rarely, occasionally, frequently or almost constantly will be used to measure anxiety and general pain. Severity of the following symptoms: Anxiety, fatigue, general pain and problems with concentration in a 7 day time period will be measured using the following scale: Mild, Moderate, Severe, Very Severe.
To quantify the change over time in PRO-CTCAE derived symptoms | Month 6 following completion of chemotherapy
  Changes in symptoms will be assessed this outcome will be measured using PRO-CTCAE Derived Symptoms and other PROs. A scale Yes or No is utilized to describe whether the following symptoms have been experienced: Anxiety, constipation, decreased appetite, diarrhea, fatigue, general pain, insomnia, mouth sores, muscle pain, nausea, numbness and tingling, problems and concentration, rash, sad, shortness of breath, vomiting. The following scale: Rarely, occasionally, frequently or almost constantly will be used to measure anxiety and general pain. Severity of the following symptoms: Anxiety, fatigue, general pain and problems with concentration in a 7 day time period will be measured using the following scale: Mild, Moderate, Severe, Very Severe.

CONTACTS AND LOCATIONS:
Overall Officials: Priya P Gor, MD, MSCE, Principal Investigator — Penn Medicine
Locations (1):
- Virtua Health, Voorhees Township, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No